CLINICAL TRIAL: NCT00858598
Title: Pro Osteon Bone Void Filler Data Collection
Brief Title: Pro Osteon Bone Void Filler Study
Acronym: PO
Status: Withdrawn | Type: Observational
Why Stopped: Study never started. Study suspended indefinitely.
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: US 6
Record Dates: First submitted 2009-03-09; First posted 2009-03-10 (Estimated); Last update posted 2017-06-21 (Actual); Status verified 2017-06

CONDITIONS: Osteoarthritis; Revision Arthroplasty
Keywords: Total Knee Arthroplasty; Revision; Tibial; Void; Bone Filler
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pro Osteon: All patients in this pilot study will receive pro osteon as a bone void filler and will be enrolled according to the same inclusion / exclusion criteria.

SUMMARY:
This study was designed to observe the outcomes of Pro Osteon according to its cleared indications for use.

DETAILED DESCRIPTION:
The purpose of this prospective clinical data-collection is to document the performance and clinical outcomes of Pro Osteon® as a Bone Void Filler. FDA has cleared this device via premarket notifications 510(k) K063346, K980817, and K990131. There will be no experimental or investigational devices used.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria will be the same as the stated indications stated in the summary of the FDA approved 510(k) K063346, K980817, and K990131 application. These indications are stated below:

* PRO OSTEON® 500R Resorbable Bone Graft Substitute is indicated only for bony voids or gaps that are not intrinsic to the stability of the bony structure.
* PRO OSTEON® 500R is indicated to be gently packed into bony voids or gaps of the skeletal system (i.e, the extremities, spine and pelvis). These defects may be surgically created osseous defects or osseous defects created from traumatic injury to the bone. PRO OSTEON® 500R can be combined with autogenous blood, and/or sterile fluids (saline or Ringer's solution). The product provides a bone void filler that resorbs and is replaced with bone during the healing process.
* Surgical techniques and patient care are to be standard for the surgeon participating in the protocol and should be maintained the same throughout the course of the data-collection.
* All patients must sign an IRB-approved Informed Consent to be enrolled into the study.

Exclusion Criteria:

Exclusion criteria will be the same as the stated contraindications stated in the summary of the FDA approved 510(k) K063346, K980817, and K990131 application. These contraindications are stated below:

* Pro Osteon® 500R Resorbable Bone Graft Substitute is contraindicated for fractures of the growth plate
* For segmental defects
* For indications which may be subjected to excessive impact or stresses
* When there is significant vascular impairment proximal to the graft site
* When there are metabolic or systemic bone disorders that affect bone or wound healing
* In infected sites
* When stabilization of the defect is not possible.
* The use of Pro Osteon® 500R is also contraindicated in cases where intraoperative soft tissue coverage is not planned or possible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who fit within the inclusion / exclusion criteria of the FDA cleared indications for use.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2009-12; Primary Completion 2013-07 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
Radiographic Evaluation | 3 Years

SECONDARY OUTCOMES:
Knee Society Score | 3 Years

REFERENCES:
- [Background] Kurtz S, Ong K, Lau E, Mowat F, Halpern M. Projections of primary and revision hip and knee arthroplasty in the United States from 2005 to 2030. J Bone Joint Surg Am. 2007 Apr;89(4):780-5. doi: 10.2106/JBJS.F.00222. PMID 17403800
- [Background] Harris AI, Poddar S, Gitelis S, Sheinkop MB, Rosenberg AG. Arthroplasty with a composite of an allograft and a prosthesis for knees with severe deficiency of bone. J Bone Joint Surg Am. 1995 Mar;77(3):373-86. doi: 10.2106/00004623-199503000-00007. PMID 7890786
- [Background] Chapman MW: Bone grafting. Chapman MW, Madison M (eds.): Operative Orthopaedics. Philadelphia, JB Lippincott, 1993, pp 139-49
- [Background] Lewonowski K, Dorr LD. Revision of cementless total knee arthroplasty with massive osteolytic lesions. J Arthroplasty. 1994 Dec;9(6):661-3. doi: 10.1016/0883-5403(94)90121-x. No abstract available. PMID 7699380
- [Background] Insall JN, Dorr LD, Scott RD, Scott WN. Rationale of the Knee Society clinical rating system. Clin Orthop Relat Res. 1989 Nov;(248):13-4. PMID 2805470
- [Background] Amstutz HC, Thomas BJ, Jinnah R, Kim W, Grogan T, Yale C. Treatment of primary osteoarthritis of the hip. A comparison of total joint and surface replacement arthroplasty. J Bone Joint Surg Am. 1984 Feb;66(2):228-41. PMID 6693450